CLINICAL TRIAL: NCT03881917
Title: Cystatin C and Beta 2 Microglobulin as Biochemical Markers for Early Detection of Renal Impairment in Children With Beta Thalassemia
Brief Title: Cystatin c and Beta 2 Microglobulin in Thalassemic Children.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Naguib Khairy, Principle Investigator, Assiut University
Other Study IDs: Renal markers in thalassemia.
Record Dates: First submitted 2019-03-18; First posted 2019-03-20 (Actual); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Blood Disease
Keywords: renal impairment
MeSH Terms: conditions — Hematologic Diseases; Renal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Cystatin c and beta 2 microglobulin kits — Kits for measurement concentration

SUMMARY:
Beta thalassemia has many complications on many systems as the renal system.So early detection of renal impairment is required in those children to decrease complications of this nephropathy.

DETAILED DESCRIPTION:
Thalassemia syndromes are the most common single gene disorders worldwide especially in developing countries. The use of regular and frequent blood transfusions in patients with beta thalassemia major has improved patients' life spans and quality of life, but can lead to chronic iron overload. Many factors contribute to the functional abnormalities found in beta thalassemia patients such as decreased red cell life span, rapid iron turnover, tissue deposition of excess iron and also, specific iron chelators can affect kidneys. The success in management of patients of beta thalassemia has led to chronic hemosiderosis in different organs like liver and heart and long-term complications in other organs like pancreas and kidneys have recently been studied. The evidence of proximal tubular damage has been observed in beta thalassemia patients. Also, low-molecular-weight proteinuria has been found in almost all patients. Unlike other organs, it is unclear whether kidney damage results solely from intravascular haemolysis, chronic transfusion or as a complication of iron chelation therapy. Although the early identification of patients at high risk of renal impairment is of great importance as it may allow specific measures to be taken to delay renal impairment, there are limited studies about renal dysfunction in pediatric thalassemic patients. Thus, in this study we will use different measurements for early detection of renal impairment even if the patients have no symptoms to handle with the disease in its reversible stage before being irreversible. Beside the usual investigations of renal function we will measure cystatin c and beta2 microglobulin as early markers of renal impairment.

ELIGIBILITY:
Inclusion Criteria:

* Children with beta thalassemia from the age of 1 year to 18 years.

Exclusion Criteria:

* Children who have other hematological or chronic disease.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children with beta thalassemia from the age of 1 year to 18 years.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-11-01 (Estimated); Primary Completion 2020-11-01 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
mean difference of cystatin c and beta 2 microglobulin concentrations with normal range | baseline
  Analysis of the results to differentiate the affected from non affected patients

REFERENCES:
- [Result] den Bakker E, Gemke RJBJ, Bokenkamp A. Endogenous markers for kidney function in children: a review. Crit Rev Clin Lab Sci. 2018 May;55(3):163-183. doi: 10.1080/10408363.2018.1427041. Epub 2018 Feb 1. PMID 29388463
- [Result] Annayev A, Karakas Z, Karaman S, Yalciner A, Yilmaz A, Emre S. Glomerular and Tubular Functions in Children and Adults with Transfusion-Dependent Thalassemia. Turk J Haematol. 2018 Mar 1;35(1):66-70. doi: 10.4274/tjh.2017.0266. Epub 2017 Jul 28. PMID 28753129
- [Result] Behairy OG, Abd Almonaem ER, Abed NT, Abdel Haiea OM, Zakaria RM, AbdEllaty RI, Asr EH, Mansour AI, Abdelrahman AM, Elhady HA. Role of serum cystatin-C and beta-2 microglobulin as early markers of renal dysfunction in children with beta thalassemia major. Int J Nephrol Renovasc Dis. 2017 Sep 11;10:261-268. doi: 10.2147/IJNRD.S142824. eCollection 2017. PMID 28979155
- [Result] Deveci B, Kurtoglu A, Kurtoglu E, Salim O, Toptas T. Documentation of renal glomerular and tubular impairment and glomerular hyperfiltration in multitransfused patients with beta thalassemia. Ann Hematol. 2016 Feb;95(3):375-81. doi: 10.1007/s00277-015-2561-2. Epub 2015 Nov 23. PMID 26596972
- [Result] Hashemieh M, Radfar M, Azarkeivan A, Hosseini Tabatabaei SMT, Nikbakht S, Yaseri M, Sheibani K. Renal Hemosiderosis among Iranian Transfusion Dependent beta-Thalassemia Major Patients. Int J Hematol Oncol Stem Cell Res. 2017 Apr 1;11(2):133-138. PMID 28875008
- [Result] Ali BA, Mahmoud AM. Frequency of glomerular dysfunction in children with Beta thalassaemia major. Sultan Qaboos Univ Med J. 2014 Feb;14(1):e88-94. doi: 10.12816/0003341. Epub 2014 Jan 27. PMID 24516760
- [Result] Bakr A, Al-Tonbary Y, Osman G, El-Ashry R. Renal complications of beta-thalassemia major in children. Am J Blood Res. 2014 Sep 5;4(1):1-6. eCollection 2014. PMID 25232499
- [Result] Uzun E, Balci YI, Yuksel S, Aral YZ, Aybek H, Akdag B. Glomerular and tubular functions in children with different forms of beta thalassemia. Ren Fail. 2015;37(9):1414-8. doi: 10.3109/0886022X.2015.1077314. Epub 2015 Sep 12. PMID 26365703
- [Result] Nickavar A, Qmarsi A, Ansari S, Zarei E. Kidney Function in Patients With Different Variants of Beta-Thalassemia. Iran J Kidney Dis. 2017 Mar;11(2):132-137. PMID 28270645